CLINICAL TRIAL: NCT05738629
Title: A Clinical Study of the Safety and Efficacy of Pluripotent Stem Cell-derived Mesenchymal Stem Cell Exosome (PSC-MSC-Exo) Eye Drops Treatment for Dry Eye Diseases Post Refractive Surgery and Associated With Blepharospasm
Brief Title: Safety and Efficacy of Pluripotent Stem Cell-derived Mesenchymal Stem Cell Exosome (PSC-MSC-Exo) Eye Drops Treatment for Dry Eye Diseases Post Refractive Surgery and Associated With Blepharospasm
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang University (Other); Hangzhou yuansheng biotechnology Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0290
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Dry Eye Disease
Keywords: dry eye disease; post refractive surgery; blepharospasm; exosomes; mesenchymal stem cell; pluripotent stem cell
MeSH Terms: conditions — Dry Eye Syndromes; Blepharospasm | interventions — Ophthalmic Solutions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PSC-MSC-Exo Eye Drops Treatment (Experimental): Participants will receive artificial tears for 2 weeks to get the normalized baseline, followed by PSC-MSC-Exo eye drop intervention for 12 weeks.
  Interventions: Drug: Pluripotent Stem Cell-derived Mesenchymal Stem Cell Exosome (PSC-MSC-Exo) Eye Drops

INTERVENTIONS:
Drug: Pluripotent Stem Cell-derived Mesenchymal Stem Cell Exosome (PSC-MSC-Exo) Eye Drops — Participants will receive artificial tears for 2 weeks to get the normalized baseline, followed by PSC-MSC-Exo eye drops 0.125 ml/single eye/one time, four times a day for 12 weeks. The follow-up visit will be 12 weeks since the administration of PSC-MSC-Exo eye drops.

SUMMARY:
The purpose of this study is to evaluate the preliminary safety and effectiveness of Pluripotent Stem Cell-derived Mesenchymal Stem Cell Exosome (PSC-MSC-Exo) Eye Drops in the treatment of dry eye diseases post refractive surgery and associated with blepharospasm

DETAILED DESCRIPTION:
Dry eye disease (DED) is a multifactorial disease of the ocular surface characterized by instability of the tear film and the prevalence has been estimated to reach 20%-40%. Especially, dry eye symptoms are common complaints of patients with blepharospasm or refractive surgery history, seriously affecting their quality of life. There are many conventional therapies for DED which include ocular lubricants, oral essential fatty acid supplementation, lid hygiene and warm compresses, punctal occlusion, various treatments to obstructed meibomian glands, topical antibiotics, topical corticosteroids, topical secretagogues, topical non-glucocorticoid immunomodulatory drugs and scleral contact lenses. However, the overall efficacy is still unsatisfactory with apparent side effects, long periods of treatment, and high-costs. Mesenchymal stem cell-derived exosomes (MSC-Exo) are 30-150nm microvesicles secreted by mesenchymal stem cells (MSCs), which can mediate the therapeutic efficacy of mesenchymal stem cells by the encapsulated proteins, miRNAs and other bioactive substances, and showed potential in the treatment of various diseases. This study aims to evaluate the preliminary safety and effectiveness of PSC-MSC-Exo in the treatment of dry eye diseases post refractive surgery and associated with blepharospasm.

This is an open-label, single-arm, before-after study with 12 subjects with dry eye diseases and the history of refractive surgery or blepharospasm. There are 5 visits over the course of 12 weeks. Visit 1: Week-1 Visit 2: Week-2 Visit 3: Week-4 Visit 4: Week-8 Visit 5: Week-12

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of apparent dry eye symptoms by ophthalmologists.
* patients experience dry eye symptoms with a definitive history of FS-LASIK or SMILE surgery, or blepharospasm, and previous application of artificial tears for more than 3 months could not relieve the dry eye symptoms.
* have the following symptoms in at least one eye: dryness, burning sensation, foreign body sensation, discomfort in the ocular surface or visual fatigue;
* tear secretion test (Schirmer's Test) of either eye ≤ 10 mm / 5 min;
* the corneal fluorescein staining score (FLCs) was more than 3 and less than 6.
* Tear break up time (TBUT) is less than 10 seconds.

Exclusion Criteria:

* Those who are allergic to any component of the drug in this study;
* Pregnant or nursing women;
* Patients with active fungal, bacterial or viral keratitis or conjunctivitis;
* have serious heart, lung, liver or kidney diseases;
* Other incurable ocular diseases before the study; such as glaucoma, uveitis, retinitis pigmentosa.
* Wearing contact lenses and unwilling to take off in the study;
* Performed ocular surgery (including cataract surgery) in recent three months;
* Enrolled in other interventional clinical studies at the same time;
* Application of eye drops that might affect the clinical study in the past 24 hours;
* Unable to complete the study according to the investigators' requirements;
* Application of eye drops other than artificial tears.
* Application of systemic medication known to reduce tear production, such as anti-anxiety drugs, antipsychotics and steroids.
* Eyelids or eyelashes anomaly.
* Serious systemic diseases.
* Refused to sign the informed consent form to participate in the experiment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Change in Ocular Surface Disease Index (OSDI) | 1 weeks, 2 weeks, 4 weeks, 8 weeks,12 weeks
  The OSDI questionnaire contains 12 questions to measure dry eye symptoms. OSDI scores range from 0 to 100. The lower the score, the more alleviation of dry eye symptoms. Compared with the baseline, a reduction of more than 10 points indicates improvement.

SECONDARY OUTCOMES:
Tear Secretion Test (Schirmer test) | 1 weeks, 2 weeks, 4 weeks, 8 weeks,12 weeks
  A paper strip is placed on the eye under the lower lid for a specified time period. The length of the strip wetted by the tears was measured in millimeters. A positive change from baseline indicates an improvement in each eye.
Tear Film Break-up Time | 1 weeks, 2 weeks, 4 weeks, 8 weeks,12 weeks
  Time required for dry spots to appear on the surface of the eye after blinking was measured in seconds. A positive change from baseline indicates improvement in each eye.
Ocular Surface Staining Score | 1 weeks, 2 weeks, 4 weeks, 8 weeks,12 weeks
  Damage of the ocular surface was measured by slit-lamp examination after staining with non-toxic fluorescein sodium. Corneal and conjunctival staining were graded as per the National Eye Institute (NEI) pictorial scale. The lower the score, the less signs of dry eye disease a patient exhibits. A negative change from baseline indicates an improvement in each eye.
Best Corrected Visual Acuity (BCVA) | 1 weeks, 2 weeks, 4 weeks, 8 weeks,12 weeks
  Whether exosomes affect visual acuity.
Conjunctiva Redness Score | 1 weeks, 2 weeks, 4 weeks, 8 weeks,12 weeks
  Conjunctival hyperemia was graded in each eye under slit-lamp magnification by assigning a score of 0 to 4 for each quadrant based on comparison to the Allergan Dry Eye Redness Scale with photographic reference where: 0=Normal, vessels of bulbar conjunctiva are easily observed; 1=Trace redness; 2=Mild redness; 3=Moderate redness; 4=Severe redness, and each score is associated with a reference photo. A negative change from baseline indicates an improvement in each eye.
Tear Meniscus Height | 1 weeks, 2 weeks, 4 weeks, 8 weeks,12 weeks
  The distance between the line of reflection along the top of the tear prism to the edge of the eyelid was measured in millimeters. A positive number change from baseline indicates improvement.
Corneal confocal microscopy | 1 weeks, 2 weeks, 4 weeks, 8 weeks,12 weeks
  The morphology, distribution and quantity of corneal nerve fibers were recorded by confocal image after LASIK and SMILE.
Meibomian gland expressibility scores | 1 weeks, 2 weeks, 4 weeks, 8 weeks,12 weeks
  Squeeze the central meibomian glands of the lower eyelid and assess the expressibility of the five central glands, where 0= All glands have meibum extruded, 1= 3-4 glands have meibum extruded, 2=1-2 glands have meibum extruded, 3=no glands have meibum extruded.
Meibomian Glands Photography | 1 weeks, 2 weeks, 4 weeks, 8 weeks,12 weeks
  The morphology, quantity and blockage of meibomian gland can be assigned a score of 0 to 3 points according to meibomian gland dropout, where 0=normal without dropout; 1=meibomian gland dropout<1/3; 2=meibomian gland dropout 1/3-2/3; 3=meibomian gland dropout >2/3. The total score of upper and lower meibomian glands is 6 points, of which Grade 0=0-1 point; Grade 1=2-3 points; Grade 2=4-5 points; Grade 3=6 points.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Ye, Doc., Study Chair — 2nd Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hanzhou, Zhejiang, China

REFERENCES:
- [Derived] Randall Harrell C, Djonov V, Volarevic A, Arsenijevic A, Volarevic V. Mesenchymal Stem Cell-Sourced Exosomes as Potentially Novel Remedies for Severe Dry Eye Disease. J Ophthalmol. 2025 Jan 10;2025:5552374. doi: 10.1155/joph/5552374. eCollection 2025. PMID 39839752